CLINICAL TRIAL: NCT02373072
Title: A Phase 1, Double Blind, Sponsor Open, Randomized, Placebo-controlled, Single Ascending Dose Study To Investigate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-06649751 In Subjects With Idiopathic Parkinson's Disease
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of PF-06649751 in Subjects With Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7601009; 2014-004389-54 (EudraCT Number)
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2017-01

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Pakinson's Disease, Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — trimethobenzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Three single doses over three periods. For each of the three periods, subjects will be crossed-over from placebo or PF-06649751. Each PF-06649751 dose is separated by at least one week.
  Interventions: Drug: PF-06649751; Drug: Trimethobenzamide Hydrochloride; Drug: Placebo
- Cohort 2 (Experimental): Three single doses over three periods. For each of the three periods, subjects will be crossed-over from placebo or PF-06649751. Each PF-06649751 dose is separated by at least one week.
  Interventions: Drug: PF-06649751; Drug: Trimethobenzamide Hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: PF-06649751 — Subjects completing all three treatment periods will be administered two doses. Doses: 0.75mg, 1.5mg, 3mg, 6mg, 9mg. Tablets in the form of 0.25mg or 1 mg.
Drug: Trimethobenzamide Hydrochloride — 300mg TID, Capsules. Optional in both Cohorts.
Drug: Placebo — Subjects completing all three treatment periods will be receiving placebo once.

SUMMARY:
This is a study with two sequential cohorts, each with three treatment periods. Single doses of PF-06649751 will be tested in this study, starting at a low dose and escalating to a dose projected to be under the current limits for drug concentration. Each cohort will aim to achieve approximately 9 completers. Primary endpoint is safety and tolerability, secondary endpoint is MDS-UPDRS part III.

ELIGIBILITY:
Inclusion Criteria:

* L-DOPA-responsiveness
* Hoehn & Yahr Stage II-III inclusive
* Experiencing motor fluctuations
* Stable daily dose of L-DOPA of at least 300 mg
* Females on non-childbearing potential and male subjects

Exclusion Criteria:

* History of troublesome dyskinesias
* History of surgical intervention for Parkinson's disease

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects with Adverse Events (AEs) | Day 1 through 61
Number of participants with vital signs data that meet criteria of potential clinical concern | Day 1 through 61
Number of participants with ECG data that meet criteria of potential clinical concern | Day 1 through 61
Number of participants with abnormal clinically significant laboratory measurements | Day 1 through 61
C-SSRS (suicidality assessment) | Day 1 through 61

SECONDARY OUTCOMES:
MDS-UPDRS part III | Day 1, Periods 1-3
  MDS - Unified Parkinson's Disease Rating Scale Part III

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (7):
  - Collaborative Neuroscience Network, LLC., Long Beach, California
  - MD Clinical, Hallandale, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland
  - Parkinson's Movement Disorder Center of Maryland, Elkridge, Maryland
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Walnut Hill Medical Center, Dallas, Texas
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Sohur US, Gray DL, Duvvuri S, Zhang Y, Thayer K, Feng G. Phase 1 Parkinson's Disease Studies Show the Dopamine D1/D5 Agonist PF-06649751 is Safe and Well Tolerated. Neurol Ther. 2018 Dec;7(2):307-319. doi: 10.1007/s40120-018-0114-z. Epub 2018 Oct 25. PMID 30361858
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7601009&StudyName=A%20Phase%201%2C%20Double%20Blind%2C%20Sponsor%20Open%2C%20Randomized%2C%20Placebo-controlled%2C%20Single%20Ascending%20Dose%20Study%20To%20Investigate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Pf-06649751%20In%20Subjects%20With%20Idiopathic%20Parkinson%E2%80%99s%20Disease